CLINICAL TRIAL: NCT02653898
Title: Defining Effective, Appropriate, Implementable Strategies for Malaria Elimination in Military Forces in Cambodia as a Model for Mobile Populations
Brief Title: Malaria Elimination Pilot Study in Military Forces in Cambodia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: National Center for Parasitology, Entomology, and Malaria Control (CNM) (Unknown); Ministry of National Defense, Royal Cambodian Armed Forces Department of Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WR2211
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Malaria; Parasitic Diseases
Keywords: Malaria; Antimalarials; Malaria Elimination; Mass Drug Administration; Malaria Prophylaxis; Mobile population; Drug resistance; Focused screening and treatment; Monthly Malaria Prophylaxis; Mass screening and treatment; Primaquine; Malaria transmission; Permethrin insecticide; Thai-Cambodian border; Cambodia; AFRIMS
MeSH Terms: conditions — Malaria; Parasitic Diseases | interventions — Primaquine; Artesunate; Mefloquine; Permethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Focused Screening and Treatment + ITU (Active Comparator): Approved antimalarial based on the malaria species identified on the monthly follow ups, following national treatment guidelines in Cambodia AND Insecticide Treated Uniform with 40% Permethrin; DHA-PIP or Artesunate + Mefloquine based on the malaria species, single dose Primaquine 15 mg in subjects with P.f uncomplicated malaria or Primaquine 45 mg weekly x 8 weeks in G6PD-deficient volunteers, or Primaquine 15 mg daily for 14 days in G6PD-normal volunteers.
  Interventions: Drug: DHA-PIP; Drug: Primaquine; Drug: Artesunate + Mefloquine; Drug: Permethrin (Insecticide treated uniform)
- Focused Screening and Treatment + sITU (Active Comparator): Approved antimalarial based on the malaria species identified at the monthly follow up and following national treatment guidelines in Cambodia AND sham treated uniform. DHA-PIP or Artesunate + Mefloquine based on the malaria species, single dose Primaquine 15 mg in subjects with P.f uncomplicated malaria or Primaquine 45 mg weekly x 8 weeks in G6PD-deficient volunteers, or Primaquine 15 mg daily for 14 days in G6PD-normal volunteers.
  Interventions: Drug: DHA-PIP; Drug: Primaquine; Drug: Artesunate + Mefloquine
- Monthly Malaria Prophylaxis + ITU (Active Comparator): Monthly DHA-PIP + weekly Primaquine 22.5 mg for 3 months; All subjects will also receive insecticide treated uniforms with 40% Permethrin
  Interventions: Drug: DHA-PIP; Drug: Primaquine; Drug: Permethrin (Insecticide treated uniform)
- Monthly Malaria Prophylaxis + sITU (Active Comparator): Monthly DHA-PIP + weekly Primaquine 22.5 mg for 3 months; All subjects will also receive sham treated uniforms
  Interventions: Drug: DHA-PIP; Drug: Primaquine

INTERVENTIONS:
Drug: DHA-PIP — Administered monthly (weight-based) on days 1-3, during months 1, 2, and 3 in the MMP arm and also as a first line agent for P.v malaria recurrence in both MMP and FSAT treatment arms
  Other Names: DHA-piperaquine; Dihydroartemisinin-piperaquine
Drug: Primaquine — 22.5 mg weekly for 12 weeks in the MMP arm; low dose primaquine (15mg) for transmission blocking of P. falciparum or 14 days of primaquine (15mg) in G6PD normal volunteers or 8 weeks of low dose primaquine (45mg) in G6PD-deficient volunteers for radical cure of P. vivax
Drug: Artesunate + Mefloquine — Weight based; first line agent for P.f malaria infection diagnosed at monthly follow ups, administered on days 1-3 in subjects with malaria recurrence
  Other Names: ASMQ; Artesunate-Mefloquine
  Arms: Focused Screening and Treatment + ITU; Focused Screening and Treatment + sITU
Drug: Permethrin (Insecticide treated uniform) — 40% Permethrin IDA kit, applied once to the uniforms for volunteers assigned to ITU arm
  Arms: Focused Screening and Treatment + ITU; Monthly Malaria Prophylaxis + ITU

SUMMARY:
Antimalarial drug resistance has reached critical levels on the Thai-Cambodian border. Many have begun advocating for concerted malaria elimination efforts in Cambodia. However, there is currently no consensus on how malaria elimination is to be achieved with the tools available.

In this study, the investigators will conduct operational research with the Royal Cambodian Armed Forces (RCAF) and National Malaria Center (CNM) to quantify the relative effectiveness of the two major interventional approaches - monthly malaria prophylaxis (MMP) or focused screening and treatment (FSAT) - in a head to-head comparison. In addition, the investigators will quantify the relative contribution of a recently advocated vector intervention for military personnel - the insecticide treated uniform (ITU) - in addition to other vector control measures currently employed by the RCAF. The investigators will employ the same permethrin insecticide self-application kits currently used by the US military. The investigators will estimate the cost effectiveness of each approach and attempt to define the best way forward for malaria elimination efforts in a critically important malaria reservoir in military population (and their dependents) who reside on the Thai-Cambodian border. The aim of the study is not only to conduct research to better define the best way forward in malaria elimination efforts in the high risk military populations, but to also build capacity within the RCAF to support and lead future elimination efforts in the most difficult-to-reach mobile populations.

DETAILED DESCRIPTION:
This is a cluster-randomized, open label interventional study to determine the feasibility of achieving significant reduction in malaria cases in military encampments on the Thai-Cambodian border. The study will compare the effectiveness, safety, and tolerability of monthly malaria prophylaxis (MMP) to monthly focused screening and treatment (FSAT). This study will thus investigate the effectiveness of two potential interventions for malaria elimination. Subjects in the monthly malaria prophylaxis (MMP) arm will receive a standard 3-day treatment course of dihydroartemisinin-piperaquine on months 1, 2 and 3 and weekly low-dose primaquine (22.5mg for 12 weeks). Volunteers in the focused screening and treatment (FSAT) arm will be screened monthly and then treated for malaria following national treatment guidelines. For G6PD-deficient volunteers in the FSAT arm, primaquine will be administered weekly (45mg for 8 weeks) as radical curative and/or presumptive anti-relapse therapy. For G6PD normal volunteers with vivax infection, primaquine will be administered daily (15mg for 14 days). All FSAT volunteers with confirmed P. falciparum infection will receive a single, low dose (15mg) Primaquine as a P. falciparum transmission-blocking agent. The incremental benefit of an insecticide treated uniform (ITU) will also be assessed as a single-blind sham-controlled intervention in addition to personal protective measures currently employed by the RCAF. Volunteers will be followed monthly for a total of 6 months, to determine the proportion remaining malaria-free on day 180 following enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Military volunteers aged 18-65 years of age plus their dependents > 2 years of age, eligible for care at an RCAF facility, or otherwise eligible Cambodian civilians at risk for contracting malaria who live within the designated geographical areas
2. Able to give informed consent/assent
3. Resides in the selected study areas, and available for monthly follow-up for 6 month study duration
4. Agrees not to seek outside medical care for febrile illness unless referred by study team
5. Authorized by local commander to participate in the study if on active duty

Exclusion Criteria:

1. Allergic reaction or contraindication to dihydroartemisinin-piperaquine or primaquine or artesunate+mefloquine
2. Pregnant or lactating female, or female of childbearing age, up to 50 years of age or otherwise individually assessed for childbearing potential, who does not agree to use an acceptable form of contraception during the study
3. Judged by the investigator to be otherwise unsuitable for study participation

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The absolute risk reduction based on the proportion of subjects remaining malaria-free at the end of 6 months between the study arms as diagnosed by PCR-corrected malaria microscopy | 6 months

SECONDARY OUTCOMES:
Overall rate of sexual stage infections at Months 1 through 6 in each arm based on a combined endpoint of light microscopy and PCR analysis for detection of gametocyte maturity. | 6 months
Number of participants with abnormal lab values and/or Adverse Events that are related to the treatments in each arm | 6 months
Kaplan-Meier survival analysis of asexual and sexual blood stage at 28-day intervals after treatment or prophylaxis up to 180 days | 6 months
Comparison of all-species and species-specific malaria incidence density in each arm over 180-day period | 6 months
Comparative incidence of malaria detected by RDT versus RT-PCR versus microscopy | 6 months
Comparative incidence of G6PD deficiency in the study population as determined by RDT, quantitative, and qualitative tests | At the time of enrollment
Estimate of apparent rates of preexisting immunity to malaria based on medical history, days of fever prior to presentation, and preexisting parasitological parameters (gametocytemia, low asexual stage parasitemias) | 6 months
Sensitivity and specificity assessment of the currently recommended rapid diagnostic test in Cambodia to detect moderate to severe G6PD deficiency using quantitative G6PD testing as the reference standard | At the time of enrollment
Odds ratio for P.v recurrence for each CYP2D6 phenotype | 6 months
Rate of cytochrome P450 2D6 genotypes/phenotypes in the population at risk | 6 months
Percent reduction in hemoglobin and HTC for each 2D6 haplotype in subjects with available CBC following PQ dosing | Day 3 (and day 7 in those volunteers with Hgb or HCT drop of at least 10% from baseline on Day 3)
Percentage of subjects with malaria recurrence for each CYP2D6 phenotype | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chanthap Lon, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand; Mariusz Wojnarski, MD, Study Chair — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (1):
- RCAF treatment facilities, Anlong Veaeng, Oddar Meancheay, Cambodia

IPD SHARING:
Plan to Share IPD: Yes
The preliminary results, final report and key data will be shared with a broad array of stakeholders from Cambodia, the region, bilateral and multilateral implementing partners, and donor organizations.

REFERENCES:
- [Derived] Manning J, Lon C, Spring M, Wojnarski M, Somethy S, Chann S, Gosi P, Soveasna K, Sriwichai S, Kuntawunginn W, Fukuda MM, Smith PL, Rekol H, Sinoun M, So M, Lin J, Satharath P, Saunders D. Cluster-randomized trial of monthly malaria prophylaxis versus focused screening and treatment: a study protocol to define malaria elimination strategies in Cambodia. Trials. 2018 Oct 16;19(1):558. doi: 10.1186/s13063-018-2931-x. PMID 30326952